CLINICAL TRIAL: NCT04301310
Title: A Phase 1, Open-label Study to Evaluate the Effect of Rifampin on the Single Dose Pharmacokinetics, Safety, and Tolerability of BMS-986235 in Healthy Participants
Brief Title: Study to Evaluate the Effect of Rifampin on the Drug Levels in Blood and Safety of BMS-986235 in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV018-023
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Drug: BMS-986235 (Treatment A); Drug: Rifampin (Treatment B)

INTERVENTIONS:
Drug: BMS-986235 (Treatment A) — Specified dose on specified days
Drug: Rifampin (Treatment B) — Specified dose on specified days

SUMMARY:
The purpose of this study is to examine the effect of rifampin on the drug levels in blood and safety of BMS-986235, when taken by healthy participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participants, as determined by no clinically significant deviation from normal in physical examination, ECGs, and clinical laboratory determinations; no significant findings in medical history.
* Body mass index of 18.0 kg/m2 to 30.0 kg/m2, inclusive, at screening
* Males must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Women of childbearing potential (WOCBP)
* Known previous exposure to BMS-986235
* History of any significant drug allergy

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of BMS-986235 | Day 1
Area under the plasma concentration-time curve from time 0 to time of last quantifiable concentration (AUC(0-T)) of BMS-986235 | Day 1
Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC(INF)) of BMS-986235 | Day 1
Cmax of BMS-986235 with rifampin | Day 10
AUC(0-T) of BMS-986235 with rifampin | Day 10
AUC(INF) of BMS-986235 with rifampin | Day 10

SECONDARY OUTCOMES:
Incidence of Nonserious Adverse Events (AEs) | Up to 46 days
Incidence of Serious Adverse Events (SAEs) | Up to 74 days
Incidence of AEs leading to discontinuation | Up to 13 days
Incidence of clinically significant changes from baseline in physical examination findings | Up to 41 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 41 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 41 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 41 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 41 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters | Up to 41 days
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 41 days
Incidence of clinically significant changes in clinical laboratory results: Clinical chemistry tests | Up to 41 days
Incidence of clinically significant changes in vital signs: Oxygen saturation (the amount of oxygen in blood (SpO2)) | Up to 41 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm